CLINICAL TRIAL: NCT04712799
Title: The Role of the Nose for Physical Capacity
Brief Title: Nasal Breathing and Physical Capacity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SorlandetHF steinsvåg
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Nasal Obstruction; Copd
Keywords: nose; lungs; physical capacity
MeSH Terms: conditions — Nasal Obstruction; Pulmonary Disease, Chronic Obstructive | interventions — xylometazoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- COPD patients (Experimental): Wlaking tests before and afrer 1 spray with oxymetazoline
  Interventions: Drug: Otrivin

INTERVENTIONS:
Drug: Otrivin — oxymetazoline nasal spray

SUMMARY:
We know that there is a link between disorders in the upper and lower airways, both epidemiologically, patho-physiologically, and therapeutically. What we know less about is the role for the nose and nasal breathing for physical capacity. That goes both for the ability of the average, healthy persons well as for patients with ie. asthma and COPD to perform daily life activities as well as exercise and for top athletes to perform their maximum oxygen demanding activities. Without this knowledge, we cannot make evidence based decisions about to what extent measures to open the nose medically and/or surgically should be considered to improve physical capacity at any level. The aim of the present project is to expand our knowledge in the field for the best of the ordinary man, patients with airway disorders, and athletes.

DETAILED DESCRIPTION:
Nasal breathing as a prerequisite for global airway health and physical capacity,

1. Introduction The airways are traditionally divided into two segments, the upper and lower. The former consists of the nose, the paranaseal sinuses, the epipharynx, the oropharynynx, and the hypopharynx down to the level of the vocal cords. The latter involves everything below the vocal cords, including the trachea, the bronchi, the bronchioles, and the alveoli. The latter is the segment where the oxygen/CO2 exchange take place, critical for life. In this way, the upper and lower airways can be considered as two of a kind ((Steinsvag 2009). The role of the nose in this is to filter, temper and humidify the inspired air before entering the lungs. Further, the nose adds nitrogen monoxide, thereby optimizing the muco-ciliary activity and the ventilation-perfusion ratio in the lungs.

   We know that there is a link between disorders in the upper and lower airways, both epidemiologically, patho-physiologically, and therapeutically (Fireman 2000, Thorstensen, Bugten et al. 2012, Bousquet, Schünemann et al. 2019, Oie, Dahlslett et al. 2020). What we know less about is the role for the nose and nasal breathing for physical capacity. That goes both for the ability of the average, healthy persons well as for patients with ie. asthma and COPD to perform daily life activities as well as exercise and for top athletes to perform their maximum oxygen demanding activities. Without this knowledge, we cannot make evidence based decisions about to what extent measures to open the nose medically and/or surgically should be considered to improve physical capacity at any level. The aim of the present project is to expand our knowledge in the field for the best of the ordinary man, patients with airway disorders, and athletes.
2. Needs description The main impact of the present project is an improved understanding of the role of the upper airways for physical capacity. Physical capacity is essential for the ability to be physically active, move around, exercise and perform sports at any level. Thus, it is essential for the general well-being for everybody, essential as a disease-preventing factor, and essential for athletes. We know that nasal obstruction has negative impact on the lower airways, sleep(Migueis, Thuler et al. 2016), taste and smell(Dileo and Amedee 1994) as well as general quality of life(Osborn and Sacks 2013). But we do not know much about how nasal obstruction affects physical capacity. It is possible to deduce that measures to reduce mucosal inflammation in the nose and to improve nasal patency may have beneficial effects. There is scientific support for this in that intranasal steroids, cromolyn, antihistamines, and decongestants(Bousquet, Schünemann et al. 2019), which provide relief of nasal symptoms in patients with both allergic rhinitis and asthma, will also improve the pulmonary symptoms in allergic asthma(Fireman 2000). Surgical management of sinonasal pathology can improve asthma(Dunlop, Scadding et al. 1999) In some studies, external nasal dilators have been shown to improve endurance (Ottaviano, Ermolao et al. 2017). However, this has been opposed by others(Adams and Peiffer 2017).

   To be able to move around is important for most people. It is important for those with severe airway limitations/disabilities to be able to carry out elementary daily life activities as well as for most top athletes in their chase for trophies. Movement presupposes physical capacity at some level, from the lowest to the most extreme. When it comes to airway limitations, the focus usually is on the lower airways while the upper airways are forgotten. Given the unified airway concept, this is unfortunate,since optimizing the latter may have major impact on the global airway function. This implies reducing inflammation by medical means and/or improving patency by medical or surgical means, i.e. turbinate surgery, septal surgery and polypectomy.

   Before involving measures on the upper airway to improve physical capacity, we need to know more about the potential. That is the motivation for this investigation. This research project may have an impact for patients, the ordinary man, and athletes where the airways may be a limiting factor for their daily life activities and self-expression.

   Hypotheses, aims and objectives

   Hypothesis: The upper airways may have major impact on the global airway and physical capacity

   Primary aims:
   * Explore physical capacity under increasing physical strain in athletes while:

     * Breathing through the mouth and nose
     * Breathing only through the nose
     * Breathing only through the mouth.
   * Explore signs and symptoms from the upper airways in athletes and controls
   * Explore the effect of measures to improve nasal patency on physical capacity in patients with COPD.

   Objectives: To be able to optimize the physical capacity in patients with lower airway diseases, ordinary people and athletes by reducing or eliminating potentially limiting factors in the upper airways.

   During the project period, we expect to obtain evidence-based knowledge about the upper airways that may be employed to improve physical.
3. Project methodology 3.1. Project arrangements, method selection and analyses 3.1.1. Project arrangements: This is a co-operate project between Depts. of Otolaryngology, Head and Neck surgery, Sørlandet Hospital and Haukeland University Hospital, Dept. of Pulmonary Medicine, Akershus University Hospital, Dept. of Otolaryngology Head and Neck surgery, Sahlgrenska Hospital, Gothenburg, Sweden, and "Idrettshøgskolan", Gothenburg, Sweden 3.1.2. Methods, selection and analyses. 3.1.2.1: Project 1. Explore physical capacity under increasing physical strain in athletes while breathing through both the mouth and the nose, breathing only through the nose and breathing only through the mouth.

   Twelve Swedish elite cyclists between 20 and 40 years will be invited to participate after informed consent. They will have a VO2 max above 65 ml/min/kg body weight. They do not suffer from any known upper airway disease such as allergic rhinitis, rhino-sinusitis, moderate to severe septal deviation, or nasal polyps. They do not have asthma or chronic obstructive pulmonary disease. They are non-smokers. They do not use any kind of topical or systemic medication, Initially, the participants perform a pre-test to establish the exact VO2 max and Vmax according to standard techniques. Nasal symptoms like obstruction and running are recorded on Visual Analogue Scales(Voutilainen, Pitkäaho et al. 2016). The nose is investigated endoscopically. Spirometry is performed(Liou and Kanner 2009). Nasal geometry and nasal airflow are measured by acoustic rhinometry and peak nasal inspiratory flow, respectively(Chin, Marcells et al. 2014), before and after decongestion with oxymetazoline nasal spray 0,5 mg/ml.

   The testing: All the participants undergo 4 sessions at the test-laboratory. Initially, there is a test session. Then there are sessions where they run with oral and nasal breathing, mouth only breathing, and nose only breathing. The order of these tests is randomized for each test person. Each session takes approx. 2 hours.

   Before the tests, the participants avoid alcohol and heavy exercise for 24 hours. They log their dietary intake and repeat this before every test. They fast the night before testing. Waking up on the test day, the study person drinks 500 ml of water. When they arrive at the test station, their undressed height and weight are recorded. Blood and urinary tests are taken. The participants are eligible if the fluid balance evaluated by urine specific weight (USG) is <1,025 (Atago, Tokyo, Japan).

   After antropometric measurements, an increasingly strenous test on a test bike with mechanical breaks is performed(Monark LT2, Varberg, Sweden). Before measuring O2 consumption and CO2 production during sub-maximal load, indirect calometric testing via an online system is performed (Jaeger Oxycon Pro, Viasys Healthcare, Germany). The exhaustion test is a socalled ramp test with increasing load until maximum. Heart rate is continuously recorded as a mean pr. minute(Polar Electro OY, Kempele, Finland). Under the test station the air temperature is 200 and the relative humidity is 40-50%.

   The described scientific methods have, for many years, been used for research in rhinology at the depts. of oto-rhin-olaryngology, head and neck surgery, Sørlandet Hospital and Sahlgrenska sjukehuset, as well as in sports medicine at "Idrettshøgskolan", Gothenburg by the investigators. They have been demonstrated to be valid for research projects like this (referanse). Necessary resources, equipment and infrastructure are readily available in Gothenburg. This includes competance in statistics. Potential risks are limited to the test situation. All participants are familiar with the test bikes. If unexpected and unlikely incidents do occur, they will be taken immediately taken care of by medical and technical expertise present at the test station.

   3.1.2.2: Project 2. Explore signs and symptoms from the upper airways in athletes and controls.

   Symptoms may observed in persons with a disease or other abnormal conditions, but normally not observed in average healthy persons. But they may also be pure subjective feelings or notions, that do not reflect any disease or dysfunction. The latter is a well known phenomenon in rhinology. Subjects may have a feeling of complete nasal obstruction to an extent that interferes with their daily life activities, while clinical investigations and objective tests do not reveal any abnormalities. Likewise, i.e. an extensive septal deviation may not give rise to a subjective feeling of nasal obstruction. We have also shown that patients with asthma experience their nasal airway differently from those without(Thorstensen, Sue-Chu et al. 2014). This turns them into mouth breathers at an earlier stage of physical strain than healthy individuals. Premature switching to oronasal breathing results in inadequate conditioning and filtering of the inspired air, with drying and cooling of the lower airways, subsequent release of inflammatory cell mediators and development of an asthmatic response and asthma chronicity.

   We have recently demonstrated that patients with COPD have more signs and symptoms from the upper airways that may limit their physical capacity than controls(Oie, Dahlslett et al. 2020). In this paper we want to explore the corresponding situation in athletes.

   We will recruit athletes from "Olympiatoppen", in collaboration with their head of research Else Marthe Lybekk.

   The controls will be age and sex matched individuals recruited from businesses near by the hospital or patients attending the hospital for other illnesses, which are thought not to affect the upper and lower airways. Those who chose to participate may have been more interested in their health than the general population, but still we regard measurements on these individuals to be representative for the general population.

   These are the tools that will be employed, see the link https://nettskjema.no/a/155806#/page/1.

   Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) (Juniper and Guyatt 1991).

   This is an interviewer and self-administered disease-specific health-related quality of life instrument that measures the functional impairments that are most troublesome to adult (17-70 years) patients as a result of their rhinitis.

   It has 7 domains. Activity limitations (3 items), sleep problems (3 items), nose symptoms (4 items), eye symptoms (4 items), non-nose/eye symptoms (7 items), practical problems (3 items), and emotional function (4 items). The response is made on a 7-point scale (0 = not impaired at all - 6 = severely impaired). Reported interclass correlation coeficient is 0.86. Cronbach's alpha is not reported. Minimally important differences are change in scores greater than 0,5.

   Sino nasal outcome test 22 (SNOT-22)(Piccirillo, Merritt et al. 2002, Hopkins, Gillett et al. 2009) It is a validated, self-administered quality of life instrument specific for symptoms of rhinosinusitis and sensitive to clinical changes. It describes the health burden of rhinosinusitis by measuring; physical problems, functional limitations and emotional consequences of CRS by asking the participants to score 22 key symptoms. These are: the need to blow the nose, sneezing, runny nose, cough, postnasal discharge, thick nasal discharge, ear fullness, dizziness, ear pain, facial pain/ pressure, difficult falling asleep, waking up at night and difficulty falling asleep. With reference to symptoms the two last weeks, the participants scored each symptom from 0-5, giving a summery score, the total SNOT-22 score Visual analogue Scales (VAS)(Grant, Aitchison et al. 1999) The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. In this project we use VAS to measure 12 sino-nasal symptoms on a 100 mm line with endpoints "never" (0) and "always" (100). The symptoms are: Nasal obstruction, nasal running, snoring, apneas during sleep, nasal running, headache, mid facial pain, sinusitis, coughing, sneezing, general health, and sense of smell. Each subject was asked to grade each symptom and condition by frequency. VAS 0-30 is defined as mild disease, >30-7o as moderate disease and VAS >70 as severe rhinosinusitis affecting the patient´s quality of life. We also use VAS-scales to score nasal function in athletes and controls,

   Self-designed questionnaire "The athlete and his nose". Together with prof. Hellgren we have designed a questionnaire focusing on the athletes type of sport, level of performance, symptoms from the nose during activity, previous medical or surgical treatment of nasal disorders All questionnaires in this project are made electronic using the technology from "Nettskjema", University of Oslo. Collecting data will be web-based, and the answers are directly imported into systems for data- and statistical- analysis.

   Statistical analysis Based on a power test prior to the study, we need at least 45 patients to discover a difference between a normal population and a study population. We wanted to discover a mean difference of at least one with two-sided test of 5 % and 80 % power. As data will probably not be normally distributed, Mann-Whitney U test will be used in paired analyses. P less than 0.05 will be considered to be statistically significant. The analyses will be done using SPSS ver. 23 (Statistical Package for Social Sciences, Chicago, USA).

   Project 3. The physical capacity in patients with COPD before and after nasal decongestion evaluated by shuttle walking tests.

   Patients with COPD have more signs and symptoms from the upper airways than controls that may limit their physical capacity (Arndal, Sørensen et al. 2020, Oie, Dahlslett et al. 2020). In this study we will investigate to what extent measures to open their nose may improve their walking capability.

   This is a collaboration project with Anne Edvardsen and Gunnar Einvik at the dept. of Respiratory Medicine, Akershus University Hospital, Norway.

   Patients will be recruited from the out-patient section, dept. of Respiratory Medicine, Akershus University Hospital after informed consent. The COPD diagnosis will be confirmed by the presence of airflow obstruction, defined as an increase in FEV1 of less than 12% and 200 ml after administration of salbutamol by inhalation and a post bronchodilator FEV1/FVC ratio of < 0. Severity of airflow obstruction will be evaluated according to the GOLD 2014 criteria(Singh, Agusti et al. 2019). Pulmonary function tests will be performed according to ERS' guidelines for spirometry (Miller, Hankinson et al. 2005) with a calibrated Medikro Pro spirometer (Medikro Oy, Kuopio, Finland). The best FEV1 of three acceptable attempts will be recorded prior to and 10 minutes after administration of 0.4 mg Salbutamol aerosol in a spacer (Ventoline, Volumatic, GlaxoSmithKline, Middlesex, UK). Predicted reference values of Crapo et al will be used(Crapo, Morris et al. 1981). In all subjects, weight and height will be recorded. They will compete self-administered questionnaires (SNOT-22) and Visual Analogue Scales on symptoms and signs from the upper airways, and undergo an interview and clinical examination with nasal endoscopy by one of the 2 doctors (ENT) committed to the study. Peak Nasal Inspiratory Flow will also be recorded. Any subject with a positive reversibility test or nasal polyps at endoscopy, and subjects with a COPD diagnosis who do not satisfy the GOLD criteria for COPD, will be excluded from the study.

   The participants will then undergo an Incremental Shuttle Walk Test (ISWT) (Brown and Wise 2007). First two cones will be placed with 10 meters apart on a flat indoor space. The participants' speed is determined by a pre-recorded metronome that gives a signal for each stride pass a cone. The test will be stopped if the participants experience symptoms like chest pain or a drop in saturation, or if they are not able to keep up the walking speed. The speed is increased by 0.17 m/s every minute, and it may last 20 minutes maximum. At the end of the test the distanced walked is calculated by the amount of laps the participants managed to perform. The participants are experiencing a learning effect if the test is performed several times. Due to this matter the participants will perform the test twice.

   The Endurance Shuttle Walk Test (ESWT) is performed with the same distance as ISWT, but in at constant walking pace. The pace is calculated as 85% of the maximum sustainable walking pace from ISWT. The participants will firstly try the field during a 2-minute warm up period. The test is conducted until the participants has to stop due to symptoms or 20 minutes has passed. Before the ESWT the participants are asked to fill out BORG-scale and VAS-scale to determine level of dyspnoea and fatigue. Their blood pressure, heart rate and saturation are measured before, during and after the walking test.

   After 20 min. rest, 1 spray with Otrivin®(Oxymetazoline 0,1 mg/ml) is administered to each nostril. The patients rest for another 5 minutes. Then PNIF is recorded once again. They put another mark on a VAS-scale for nasal obstruction without being able to see the first one.

   Then the ESWT is repeated.

   3.3. Participants, organization and collaborations

   The study involves the following participants:

   Fride Uthaug Reite. Medical student and PhD-candidate. Oslo, Norway Sverre K. Steinsvåg. ENT-specialist. Senior Consultant and Professor at the Depts of Otolaryngology, Head and Neck Surgery, Sørlandet Hospital, Kristiansand and Haukeland University Hospital, Bergen, Norway. Initiator and main supervisor for Fride Reite.

   Johan Hellgren. ENT-specialist. Senior Consultant and Professor, ÖNH-kliniken, Sahlgrenska Sjukhuset, Gøteborg, Sverige. Investigator and assistant supervisor for Fride Reite.

   Mats Børjeson, MD PhD. Professor. Sahlgrenska Sjukhuset and Centrum för hälsa och prestationsutveckling, Gøteborg, Sverige. Investigator.

   Stefan Pettersson, PhD, Department of Food and Nutrition, and Sport and Science, University of Gothenburg, Investigator.

   Fredrik Edin. PhD. Department of Food and Nutrition, and Sport Science, University, of Gothenburg, Investigator. Centrum för hälsa och prestationsutveckling, Göteborg . Investigator.

   This is a collaboration project between institutions in Norway and Sweden. The research group consists of experienced investigators. Its totale competence in airway - and sports medicine ensures a successful completion of Fride Uthaug Reite's PhD.

   3.5. Plan for activities, visibility and dissemination Application to Regional Committees for Medical and Health Research Ethics (REC) in Norway and Sweden have already been submitted, application 134609/2020 (Norway).

   The complete research group will meet in Gothenburg, Sweden Oct. 3rd to set the plans for the first test sessions for the athletes. Alternatively, there will be a skype-meeting that day, depending on the COVID-19 situation.

   Questionnaires about physical activity and airway health will be distributed to athletes and controls during Oct. -20.

   Patients with COPD will be tested in Jan. 2021. 3.6. Plan for implementation As soon as we learn more about the role of the nose for physical capacity, we will start to test the effect of nose-opening procedures. These are primarily medical, i.e. topical nasal decongestants and topical nasal steroids. In the case of structural reasons for nasal obstruction, these may be corrected surgically. We expect to start experiments with measures to improve nasal patency in succeeding projects, in 2021.
4. Ethical considerations We cannot see any ethical concerns about testing individuals voluntarily for the nasal contribution to their physical capacity. The testing as such does imply very limiteted risk, and medical and technical personnel will always be present at the test sites in case of any unexpected incidents.

Ethical considerations may potentially arise when the test results are to be used practically.

If the testing demonstrates a positive impact of nasal breathing on physical capacity, medical or surgical measures to improve nasal patency may also improve the capacity. This may be particularly interesting for athletes and sports medicine. If this happens to be the case an ethical debate is necessary in the perspective of doping.

.

ELIGIBILITY:
Inclusion Criteria:

COPD-

Exclusion Criteria:

* Other pulmonary diseases pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2024-01-13 (Estimated); Study Completion 2024-01-13 (Estimated)

PRIMARY OUTCOMES:
increased walking distance | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: sverre steinsvåg, MD, PhD, Principal Investigator — senior consultant, professor, investigator
Locations (1):
- Sørlandet Hospital, Kristiansand, Agder, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arndal E, Sorensen AL, Lapperre TS, Said N, Trampedach C, Aanaes K, Alanin MC, Christensen KB, Backer V, von Buchwald C. Chronic rhinosinusitis in COPD: A prevalent but unrecognized comorbidity impacting health related quality of life. Respir Med. 2020 Sep;171:106092. doi: 10.1016/j.rmed.2020.106092. Epub 2020 Aug 12. PMID 32846336
- [Background] Bousquet JJ, Schunemann HJ, Togias A, Erhola M, Hellings PW, Zuberbier T, Agache I, Ansotegui IJ, Anto JM, Bachert C, Becker S, Bedolla-Barajas M, Bewick M, Bosnic-Anticevich S, Bosse I, Boulet LP, Bourrez JM, Brusselle G, Chavannes N, Costa E, Cruz AA, Czarlewski W, Fokkens WJ, Fonseca JA, Gaga M, Haahtela T, Illario M, Klimek L, Kuna P, Kvedariene V, Le LTT, Larenas-Linnemann D, Laune D, Lourenco OM, Menditto E, Mullol J, Okamoto Y, Papadopoulos N, Pham-Thi N, Picard R, Pinnock H, Roche N, Roller-Wirnsberger RE, Rolland C, Samolinski B, Sheikh A, Toppila-Salmi S, Tsiligianni I, Valiulis A, Valovirta E, Vasankari T, Ventura MT, Walker S, Williams S, Akdis CA, Annesi-Maesano I, Arnavielhe S, Basagana X, Bateman E, Bedbrook A, Bennoor KS, Benveniste S, Bergmann KC, Bialek S, Billo N, Bindslev-Jensen C, Bjermer L, Blain H, Bonini M, Bonniaud P, Bouchard J, Briedis V, Brightling CE, Brozek J, Buhl R, Buonaiuto R, Canonica GW, Cardona V, Carriazo AM, Carr W, Cartier C, Casale T, Cecchi L, Cepeda Sarabia AM, Chkhartishvili E, Chu DK, Cingi C, Colgan E, de Sousa JC, Courbis AL, Custovic A, Cvetkosvki B, D'Amato G, da Silva J, Dantas C, Dokic D, Dauvilliers Y, Dedeu A, De Feo G, Devillier P, Di Capua S, Dykewickz M, Dubakiene R, Ebisawa M, El-Gamal Y, Eller E, Emuzyte R, Farrell J, Fink-Wagner A, Fiocchi A, Fontaine JF, Gemicioglu B, Schmid-Grendelmeir P, Gamkrelidze A, Garcia-Aymerich J, Gomez M, Gonzalez Diaz S, Gotua M, Guldemond NA, Guzman MA, Hajjam J, O'B Hourihane J, Humbert M, Iaccarino G, Ierodiakonou D, Illario M, Ivancevich JC, Joos G, Jung KS, Jutel M, Kaidashev I, Kalayci O, Kardas P, Keil T, Khaitov M, Khaltaev N, Kleine-Tebbe J, Kowalski ML, Kritikos V, Kull I, Leonardini L, Lieberman P, Lipworth B, Lodrup Carlsen KC, Loureiro CC, Louis R, Mair A, Marien G, Mahboub B, Malva J, Manning P, De Manuel Keenoy E, Marshall GD, Masjedi MR, Maspero JF, Mathieu-Dupas E, Matricardi PM, Melen E, Melo-Gomes E, Meltzer EO, Menditto E, Mercier J, Miculinic N, Mihaltan F, Milenkovic B, Moda G, Mogica-Martinez MD, Mohammad Y, Montefort S, Monti R, Morais-Almeida M, Mosges R, Munter L, Muraro A, Murray R, Naclerio R, Napoli L, Namazova-Baranova L, Neffen H, Nekam K, Neou A, Novellino E, Nyembue D, O'Hehir R, Ohta K, Okubo K, Onorato G, Ouedraogo S, Pali-Scholl I, Palkonen S, Panzner P, Park HS, Pepin JL, Pereira AM, Pfaar O, Paulino E, Phillips J, Picard R, Plavec D, Popov TA, Portejoie F, Price D, Prokopakis EP, Pugin B, Raciborski F, Rajabian-Soderlund R, Reitsma S, Rodo X, Romano A, Rosario N, Rottem M, Ryan D, Salimaki J, Sanchez-Borges MM, Sisul JC, Sole D, Somekh D, Sooronbaev T, Sova M, Spranger O, Stellato C, Stelmach R, Suppli Ulrik C, Thibaudon M, To T, Todo-Bom A, Tomazic PV, Valero AA, Valenta R, Valentin-Rostan M, van der Kleij R, Vandenplas O, Vezzani G, Viart F, Viegi G, Wallace D, Wagenmann M, Wang Y, Waserman S, Wickman M, Williams DM, Wong G, Wroczynski P, Yiallouros PK, Yorgancioglu A, Yusuf OM, Zar HJ, Zeng S, Zernotti M, Zhang L, Zhong NS, Zidarn M; ARIA Study Group; MASK Study Group. Next-generation ARIA care pathways for rhinitis and asthma: a model for multimorbid chronic diseases. Clin Transl Allergy. 2019 Sep 9;9:44. doi: 10.1186/s13601-019-0279-2. eCollection 2019. PMID 31516692
- [Background] Crapo RO, Morris AH, Gardner RM. Reference spirometric values using techniques and equipment that meet ATS recommendations. Am Rev Respir Dis. 1981 Jun;123(6):659-64. doi: 10.1164/arrd.1981.123.6.659. PMID 7271065
- [Background] Dileo MD, Amedee RG. Disorders of taste and smell. J La State Med Soc. 1994 Oct;146(10):433-7. PMID 7798776
- [Background] Dunlop G, Scadding GK, Lund VJ. The effect of endoscopic sinus surgery on asthma: management of patients with chronic rhinosinusitis, nasal polyposis, and asthma. Am J Rhinol. 1999 Jul-Aug;13(4):261-5. doi: 10.2500/105065899782102809. PMID 10485011
- [Background] Enright PL. The six-minute walk test. Respir Care. 2003 Aug;48(8):783-5. PMID 12890299
- [Background] Fireman P. Rhinitis and asthma connection: management of coexisting upper airway allergic diseases and asthma. Allergy Asthma Proc. 2000 Jan-Feb;21(1):45-54. doi: 10.2500/108854100778248935. PMID 10748952
- [Background] Fisher LH, Davies MJ, Craig TJ. Nasal obstruction, the airway, and the athlete. Clin Rev Allergy Immunol. 2005 Oct;29(2):151-8. doi: 10.1385/CRIAI:29:2:151. PMID 16251769
- [Background] Grant S, Aitchison T, Henderson E, Christie J, Zare S, McMurray J, Dargie H. A comparison of the reproducibility and the sensitivity to change of visual analogue scales, Borg scales, and Likert scales in normal subjects during submaximal exercise. Chest. 1999 Nov;116(5):1208-17. doi: 10.1378/chest.116.5.1208. PMID 10559077
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277
- [Background] Liou TG, Kanner RE. Spirometry. Clin Rev Allergy Immunol. 2009 Dec;37(3):137-52. doi: 10.1007/s12016-009-8128-z. Epub 2009 Apr 4. PMID 19347610
- [Background] Migueis DP, Thuler LC, Lemes LN, Moreira CS, Joffily L, Araujo-Melo MH. Systematic review: the influence of nasal obstruction on sleep apnea. Braz J Otorhinolaryngol. 2016 Mar-Apr;82(2):223-31. doi: 10.1016/j.bjorl.2015.05.018. Epub 2016 Jan 7. PMID 26830959
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Oie MR, Dahlslett SB, Sue-Chu M, Helvik AS, Steinsvag SK, Thorstensen WM. Rhinosinusitis without nasal polyps in COPD. ERJ Open Res. 2020 Jul 6;6(2):00015-2020. doi: 10.1183/23120541.00015-2020. eCollection 2020 Apr. PMID 32665943
- [Background] Osborn JL, Sacks R. Chapter 2: Nasal obstruction. Am J Rhinol Allergy. 2013 May-Jun;27 Suppl 1:S7-8. doi: 10.2500/ajra.2013.27.3889. PMID 23711030
- [Background] Ottaviano G, Ermolao A, Nardello E, Muci F, Favero V, Zaccaria M, Favero L. Breathing parameters associated to two different external nasal dilator strips in endurance athletes. Auris Nasus Larynx. 2017 Dec;44(6):713-718. doi: 10.1016/j.anl.2017.01.006. Epub 2017 Jan 30. PMID 28153693
- [Background] Piccirillo JF, Merritt MG Jr, Richards ML. Psychometric and clinimetric validity of the 20-Item Sino-Nasal Outcome Test (SNOT-20). Otolaryngol Head Neck Surg. 2002 Jan;126(1):41-7. doi: 10.1067/mhn.2002.121022. PMID 11821764
- [Background] Silvers WS, Poole JA. Exercise-induced rhinitis: a common disorder that adversely affects allergic and nonallergic athletes. Ann Allergy Asthma Immunol. 2006 Feb;96(2):334-40. doi: 10.1016/S1081-1206(10)61244-6. PMID 16498856
- [Background] Singh D, Agusti A, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Criner GJ, Frith P, Halpin DMG, Han M, Lopez Varela MV, Martinez F, Montes de Oca M, Papi A, Pavord ID, Roche N, Sin DD, Stockley R, Vestbo J, Wedzicha JA, Vogelmeier C. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease: the GOLD science committee report 2019. Eur Respir J. 2019 May 18;53(5):1900164. doi: 10.1183/13993003.00164-2019. Print 2019 May. PMID 30846476
- [Background] Thorstensen WM, Bugten V, Sue-Chu M, Fossland NP, Romundstad PR, Steinsvag SK. Sino-nasal characteristics in asthmatic patients. Otolaryngol Head Neck Surg. 2012 Nov;147(5):950-7. doi: 10.1177/0194599812451408. Epub 2012 Jun 19. PMID 22714421
- [Background] Voutilainen A, Pitkaaho T, Kvist T, Vehvilainen-Julkunen K. How to ask about patient satisfaction? The visual analogue scale is less vulnerable to confounding factors and ceiling effect than a symmetric Likert scale. J Adv Nurs. 2016 Apr;72(4):946-57. doi: 10.1111/jan.12875. Epub 2015 Dec 22. PMID 26689434
- [Background] Walker A, Surda P, Rossiter M, Little S. Nasal function and dysfunction in exercise. J Laryngol Otol. 2016 May;130(5):431-4. doi: 10.1017/S0022215116000128. PMID 27095550
- [Result] Steinsvag SK. [Nose and lungs--two of a kind]. Tidsskr Nor Laegeforen. 2009 Oct 8;129(19):1982-4. doi: 10.4045/tidsskr.08.0394. Norwegian. PMID 19823201